CLINICAL TRIAL: NCT02196467
Title: Transplantation of Myoblasts to Duchenne Muscular Dystrophy (DMD) Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIRUL 104501; 299825 (Other Grant/Funding Number: CIHR/IRSC)
Record Dates: First submitted 2014-05-09; First posted 2014-07-22 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: myoblast; transplantation; strength; tacrolimus; immunosuppression
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Myoblast transplantation & strength (Experimental): 30 million myoblasts will be transplanted per centimeter cube in the Extensor carpi radialis of one of the patient's forearms, resuspended in saline. The strength will be evaluated after 3 and 6 months and the presence of dystrophin after 3 or 6 months.
  Interventions: Biological: Myoblast transplantation
- Saline injection & strength (Sham Comparator): The same saline solution used in the previous arm, but without cells, will be injected similarly per centimeter cube in the Extensor carpi radialis of the contralateral patient's forearm. The strength will be evaluated after 3 and 6 months and the presence of dystrophin after 3 or 6 months.
  Interventions: Procedure: Saline injection

INTERVENTIONS:
Biological: Myoblast transplantation — 30 million myoblasts will be transplanted per centimeter cube in the Extensor carpi radialis of one of the patient's forearm, resuspended in saline (a total of 0.5 ml of suspension per centimetre cube of muscle).
  Arms: Myoblast transplantation & strength
Procedure: Saline injection — A saline solution (the same used to resuspend de myoblasts in the first intervention) will be injected similarly in the Extensor carpi radialis of the contralateral patient's forearm (a total of 0.5 ml of saline per centimetre cube of muscle).
  Arms: Saline injection & strength

SUMMARY:
This Phase I/II of the clinical trial is to investigate whether the transplantation of normal myoblasts throughout one muscle (the extensor carpi radialis) of the patients is safe and will improve the strength of that muscle. During this Phase I/II, the patients will be transplanted with myoblasts grown from the muscle biopsy of a donor and kept frozen in liquid nitrogen. Thirty million myoblasts will be injected per cm cube in a progressively higher surface of the radialis (i.e., 3, 6 and 9 cm2). The contralateral muscle will be injected with saline to serve as a control. The strength of both muscles will be measured at 3 months post transplantation to verify whether the myoblast transplantation improved the strength of the muscle. If there is no significant strength improvement, the protocol will be terminated immediately for that patient. If there is a significant strength improvement, the patient will be maintained under immunosuppression until 6 months post transplant and his strength will be re-evaluated.

DETAILED DESCRIPTION:
Duchenne Muscular Dystrophy (DMD) is a degenerative disease of genetic origin, due to a mutation in the gene coding for the protein dystrophin. This mutation leads to deficiency of dystrophin in the myofibers, causing progressive muscle degeneration by the following mechanism: (1) dystrophin deficiency leads to myofibers being very vulnerable to muscle contraction-relaxation, causing frequent damage and necrosis of myofibers; (2) necrosis is followed by myofiber regeneration, as long as the regenerative capacity of muscle is not exhausted; (3) when the regenerative capacity of the muscle is exhausted, myofibers become atrophic and are ultimately lost; (4) fibrosis and fat infiltration replace the lost myofibers. This progressive muscle destruction takes place in most muscles of the limbs and trunk, leading to progressive loss of muscle strength, musculotendinous contractures, restrictive respiratory insufficiency and premature death between 17 and 30 years.

The transplantation of myoblasts obtained from a healthy donor is a potential treatment of DMD. Following intramuscular injection, donor myoblasts fuse with the myofibers of the patient, introducing the normal dystrophin gene in them. In a previous Phase 1A clinical trial, the investigators proved that transplantation of myoblasts grown from the muscle biopsy of a healthy donor introduced the normal dystrophin gene in the DMD myofibers, with the consequent expression of the normal dystrophin mRNA and restoration of the dystrophin protein in several myofibers.

The aim of this Phase I/II of the clinical trial is to investigate whether the transplantation of normal myoblasts throughout one muscle (in this case, the extensor carpi radialis) of DMD patients is safe and will improve the strength of that muscle. The patients will be transplanted with myoblasts grown from the muscle biopsy of a healthy donor. Thirty million myoblasts will be injected per cm cube in a progressively higher volume of muscle (i.e., 3, 6 and 9 cm cube). The contralateral muscle will be injected with saline as a control. The patients and the investigators will be blind to the side injected with cells. The strength of both muscles will be measured at 3 months post transplant to verify if myoblast transplantation increased muscle strength. If there is no significant strength increase, the protocol will be terminated immediately for that patient. If there is a significant strength increase, the patient will be maintained under immunosuppression until 6 months and the muscle strength will be re-evaluated.

The objectives of this Phase I/II clinical trial with DMD patients are thus:

Primary objective:

To evaluate the safety of a procedure of high-density injections of donor myoblasts throughout a muscle (under immunosuppression by tacrolimus).

Secondary objectives:

1. To evaluate whether myoblast transplantation resulted in the presence of dystrophin-positive myofibers of donor origin.
2. To evaluate whether myoblast transplantation improved the muscle strength or prevent or slowed down the progression of the muscle weakness as shown by the following parameters:

   2.1) Increase of the voluntary strength of the subject's wrist extension done by the extensor carpi radialis 12 or 24 weeks after myoblast transplantation compared with the pre-transplant values of the same muscle.

   2.2) Reduction of the fatigue of the voluntary strength of the subject's wrist extension done by the extensor carpi radialis 12 or 24 weeks after myoblast transplantation compared with the pre-transplant fatigue values of the same muscle.

   2.3) Reduce the progression of the muscle weakness in the myoblast injected muscle compared with the control contralateral muscle.
3. To verify the long term effectiveness of the tacrolimus immunosuppression to control acute rejection in myoblast transplantation (by examining the presence of muscle fibers expressing normal dystrophin and the absence of specific immune responses)

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of DMD must be confirmed (i.e., with supporting confirmation demonstrated by the identification of a mutation in the dystrophin gene compatible with DMD or presence of less than 10% dystrophin positive fibers in a muscle biopsy in a subject with DMD).
* The subject has to be older than 16 years of age.
* Male
* If on corticosteroids, a stable dose must be maintained for 6 months prior to myoblast transplantation and throughout the trial
* A potential haplotype compatible donor (the father, the mother, a brother or sister who is more than 18 years old) should be available.
* The subject must be able to move both wrists, with an MRC scale score of greater than or equal to 2.
* Subject must have been vaccinated for pneumococcus and Haemophilus influenzae.
* For subjects who are sexually active, willingness to abstain from sexual intercourse or employ a barrier or medical method of contraception for the duration of the study.
* For subjects that need assisted ventilation, a stable regimen of non-invasive ventilation parameters for 3 months prior to the first myoblast transplantation and anticipation that they will be on a stable regimen throughout the study.
* Written informed consent of the subject and donor.

Exclusion Criteria:

* An abnormal sensory examination
* Persisting abnormal values in a hemogram (red blood cells, white blood cells, hemoglobin or platelets out of laboratory normal range).
* A history of chronic infection.
* Abnormal glycosylated hemoglobin level and/or fasting blood glucose (values out of laboratory normal range)
* Previous neoplasia.
* Previous tuberculosis or potential carrier of latent tuberculosis.
* Any clinically significant cardiac, endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease as determined by the Investigator that is not related to DMD
* Previous history of renal problems or laboratory analyses suggestive of a renal problem (cystatin C, blood urea nitrogen, electrolytes out of laboratory normal range).
* Previous biopsies or intramuscular injections in any of the extensor carpi radialis.
* Subject who participated to phase 1A of myoblast transplantation
* The subject uses a drug that is not compatible with tacrolimus (see section 6 "Concomitant medications" of protocol) within the last month. If the subject has previously used one of these drugs, the washout period before the onset of tacrolimus should be at least 1 month.
* Subject tests positive for HIV-1, HIV-2, antigen HIV-1, HBC (hepatitis B surface antigen (HBsAg) and hepatitis B core antigen) HCV, HTLV-1 and anti-HTLV-2.
* The subject was submitted to electromyography in the extensor carpi radialis, within the last 6 months.
* There are pre-existing antibodies in the subject serum against the donor lymphocytes.
* Any change (initiation, dose adjustment, interruption or discontinuation) in any medication that may affect muscle function (eg. Losartan, coenzyme Q10, green tea extract, idebenone, creatine, nutritional supplements, etc.) within 3 months of the first myoblast transplantation.
* Any change in cardiac medications (ACE inhibitor, beta-blocker, etc.) within 3 months of first myoblast transplantation.
* Any surgery or fracture of the upper extremity within 3 months prior to first myoblast transplantation or plans to have surgery during the course of the trial.
* No haplotype compatible donor is available.
* Unwillingness or inability of the subject to understand and comply with the requirements of this protocol in the opinion of the Investigator or sponsor.
* Previous tuberculosis or potential carrier of latent tuberculosis.
* Previous treatment with any other investigational product within 6 months of myoblast transplantation.

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-05; Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events as a measure of safety. | Up to 6 months
  The patients will be monitored for local and systemic potential adverse effects due to the transplantation and for adverse effects associated with immunosuppression with tacrolimus.

SECONDARY OUTCOMES:
Percentage of dystrophin-positive fibers in a muscle biopsy 3 or 6 months after myoblast transplantation. | 6 months after the myoblast transplantation
  The presence of dystrophin positive fibers will be assessed in a muscle biopsy done 6 months after the myoblast transplantation.
Strength of the Extensor carpi radialis muscles. | At 3 and 6 months after myoblast transplantation.
  The strength of both Extensor carpi radialis will be evaluated 3 and 6 months after the myoblast transplantation to evaluate whether this transplantation improved the muscle strength, prevented or slowed down the progression of the muscle weakness.
Presence of a cellular and humoral reaction against the donor antigens | Every 4 weeks after transplantation for 6 months
  To assess antibody-mediated immune responses, a blood sample will be obtained at days D-14 and D15, at week 4 and every 4 weeks until the end of the treatment schedule according to the transplant pattern of the subject, and at the 3 and 6 month follow ups. These blood samples will be used to make cross-matches to determine whether the subject is producing antibodies reacting with the donor myoblasts. The antibodies against donor myoblasts will be detected by flow cytometry. Antibodies against donor HLA class I and II antigens will also be assessed by flow cytometry using single HLA antigen-coated beads (Flow PRA beads, One Lambda, Canoga Park, CA).

CONTACTS AND LOCATIONS:
Overall Officials: Craig Campbell, MD MSc FRCPC, Principal Investigator — University of Western Ontario, Canada; Jack Puymirat, MD, Principal Investigator — Centre de recherche du CHU de Quebec
Locations (2):
- Canada (2):
  - Children's Hospital London Health Sciences Centre, London, Ontario
  - Centre de recherche du CHU de Quebec - CHUL, Québec

IPD SHARING:
Plan to Share IPD: Yes
The clinical trial results that have a relation to its objectives will be published as scientific papers in scientific journals or presented at scientific meetings, but without revealing the identity of the participants who will always remain anonymous.
Time Frame: The data will begin to be available as of the fall of 2019, not being decided yet for how long.
Access Criteria: Information to be shared will be the expression of dystrophin, changes in strength, and evidence or not of rejection, in the muscles injected, as well as the side effects observed.

REFERENCES:
- [Background] Skuk D, Goulet M, Roy B, Piette V, Cote CH, Chapdelaine P, Hogrel JY, Paradis M, Bouchard JP, Sylvain M, Lachance JG, Tremblay JP. First test of a "high-density injection" protocol for myogenic cell transplantation throughout large volumes of muscles in a Duchenne muscular dystrophy patient: eighteen months follow-up. Neuromuscul Disord. 2007 Jan;17(1):38-46. doi: 10.1016/j.nmd.2006.10.003. Epub 2006 Dec 4. PMID 17142039
- [Background] Skuk D, Goulet M, Roy B, Chapdelaine P, Bouchard JP, Roy R, Dugre FJ, Sylvain M, Lachance JG, Deschenes L, Senay H, Tremblay JP. Dystrophin expression in muscles of duchenne muscular dystrophy patients after high-density injections of normal myogenic cells. J Neuropathol Exp Neurol. 2006 Apr;65(4):371-86. doi: 10.1097/01.jnen.0000218443.45782.81. PMID 16691118
- [Background] Skuk D, Vilquin JT, Tremblay JP. Experimental and therapeutic approaches to muscular dystrophies. Curr Opin Neurol. 2002 Oct;15(5):563-9. doi: 10.1097/00019052-200210000-00007. PMID 12352000
- [Background] Hogrel JY, Zagnoli F, Canal A, Fraysse B, Bouchard JP, Skuk D, Fardeau M, Tremblay JP. Assessment of a symptomatic Duchenne muscular dystrophy carrier 20 years after myoblast transplantation from her asymptomatic identical twin sister. Neuromuscul Disord. 2013 Jul;23(7):575-9. doi: 10.1016/j.nmd.2013.04.007. Epub 2013 May 31. PMID 23731976